CLINICAL TRIAL: NCT04984473
Title: Combined Cardiac Rehabilitation and Inspiratory Muscle Training in Heart Failure
Brief Title: A Study to Evaluate Breathing Muscle Training in Cardiac Rehab
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joshua R. Smith, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20-009490
Record Dates: First submitted 2021-06-14; First posted 2021-07-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Healthy; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham arm (Sham Comparator): Perform inspiratory muscle training at 2% maximal inspiratory pressure for 12 weeks.
  Interventions: Device: Inspiratory muscle training
- Non-sham arm (Active Comparator): Perform inspiratory muscle training at 40% maximal inspiratory pressure for 12 weeks.
  Interventions: Device: Inspiratory muscle training

INTERVENTIONS:
Device: Inspiratory muscle training — Inspiratory muscle training for 12 weeks at 40% maximal inspiratory pressure

SUMMARY:
The purpose of this study is to understand if breathing muscle training combined with cardiac rehabilitation influences the blood flow and blood pressure response during exercise.

ELIGIBILITY:
Inclusion Criteria - Heart Failure Group:

* Adult 18 years and older.
* English speaking.
* Has a qualifying heart failure indication for center-based cardiac rehabilitation.

Inclusion Criteria - Healthy Control Group:

* Adult 18 years and older.
* English speaking.
* Absence of pulmonary, cardiovascular, musculoskeletal, neurologic, or orthopedic diseases. Controls will be matched for age and sex.

Exclusion Criteria:

* HF patients who are unable to engage in a regularly structured exercise training program as part of a clinically indicated center-based outpatient cardiac rehabilitation program.
* Participants unable/unwilling to provide informed consent.
* Uremia, history of allergy to iodides. Impaired renal function.
* Creatinine value greater than 1.3 mg/dL (via clinical record within the past 6 months).
* Diagnosis of liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Blood pressure response | baseline and 12 week follow up
  Mean arterial pressure
Change in blood flow response | baseline and 12 week follow up
  respiratory muscle blood flow
Change in limb vascular resistance response | baseline and 12 week follow up
  Limb vascular resistance

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Smith, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials